CLINICAL TRIAL: NCT05451368
Title: Characteristics of Intimal and Neoatherosclerosis in Patients With Restenosis After DES Implantation for Calcified Lesions
Brief Title: Neointimal Features in Patients With Restenosis of Calcified Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Zhen Fang, clinical doctor, Shenyang Northern Hospital
Other Study IDs: plz333333
Record Dates: First submitted 2022-06-21; First posted 2022-07-11 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Coronary Artery Calcification; Restenosis; Neointima; Neoatherosclerosis
Keywords: coronary artery calcification; ISR; neoatherosclerosis
MeSH Terms: conditions — Neointima

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- calcified group: A calcified coronary culprit lesion was defined as "readily apparent densities noted within the apparent vascular wall at the site of the stenosis". target lesions were classified as severe ("radio opacities noted without cardiac motion prior to contrast injection generally involving both sides of the arterial wall"),moderate ("densities noted only during the cardiac cycle prior to contrast injection").Severe and moderate calcification is classified as a calcified group.
  Interventions: Other: Coronary artery calcification lesions
- non-calcified group: none/mild(lesions other than severe and moderate calcified lesions). none/mild calcification is classified as a non-calcified group.

INTERVENTIONS:
Other: Coronary artery calcification lesions — Calcification of atherosclerosis, a complex, organic, regulated and active process, is one of the manifestations of atherosclerosis. The progression of coronary atherosclerosis is a strong independent predictor of future coronary events. It has been shown that coronary artery calcification affects the healing of the neointima and the function of the endothelium after stenting. This may lead to changes in neointimal morphology and the development of neoatherosclerosis after stent implantation.
  Groups: calcified group

SUMMARY:
Previous studies have suggested that restenosis (RS) after stenting is mainly due to smooth muscle cell proliferation and migration, but recent evidence suggests that in-stent restenosis（ISR） is associated with a number of factors. Coronary artery calcification is an independent predictor of ischaemia-mediated revascularisation 1 year after percutaneous coronary intervention (PCI) following RS.The characteristics of new neointima in patients with in-stent restenosis of calcified lesions are important issues to explore

DETAILED DESCRIPTION:
The characteristics of the endothelium after DES following implantation of calcified lesions have always been of interest to us. Its inherent peculiarities make the new endothelium of calcified lesions different.

Firstly, the presence of calcification makes the neointima heal slowly. In addition DES has an anti-proliferative effect, which further diminishes the healing ability of the neointima of calcified lesions and impairs the barrier function of the endothelium. This may have a similar pathway to the formation of neointimal atherosclerosis or heterogeneous endothelium within the neointima.

Secondly, stents with calcified lesions can be accompanied by incomplete stent expansion, stent fracture and stent misalignment. These conditions may accelerate the occurrence of restenosis within the stent.

Thirdly, there are different types of calcified lesions. Different types of calcified lesions may heal and restenosis in different ways.

It is therefore understood that calcified lesion healing has a number of pathways that exist in contradiction. These are issues that need to be explored in depth.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is older than 18 years.
2. The patient had undergone coronary angiography at our hospital for PCI and had first ISR with drug-eluting stent implantation.
3. Calcified lesion greater than 5 mm in length.
4. Stent implantation time greater than 30 days.

Exclusion Criteria:

1. Bridge vessel lesions following coronary artery bypass grafting.
2. Planned modification of the DAPT regimen for medical reasons or other surgical procedures requiring modification within 3 months of the index procedure.
3. Patients undergoing heart transplantation.
4. Significant angiogenic lesions in the target vessel that may prevent stent delivery and deployment.
5. Bifurcation disease lesions involving collateral branches ≥ 2.5 mm in diameter.
6. Lesions deemed by the investigator to be unsuitable for OCT imaging (e.g., extremely curved, very distal lesions).
7. Serum creatinine > 2.0 mg/dl at the time of treatment.
8. Greater than three types of stent implantation.
9. Subjects with malignancy or other co-morbidities (i.e., severe liver, kidney, lung, or pancreatic disease with a life expectancy of less than 18 months or which may result in protocol non-compliance).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who had previously undergone stenting in our department were first found to have restenosis due to symptomatic admission angiography, and patients with restenosis were divided into calcified and non-calcified groups according to their first coronary angiography images by OCT.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-03-17 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Mean lumen area | through study completion, an average of 1 year
  Quantitative Indicators，the mean area bounded by the luminal border on OCT（Optical Coherence Tomography）
Minimum lumen area | through study completion, an average of 1 year
  Quantitative Indicators，the minimum area bounded by the luminal border on OCT
Maximum lumen area | through study completion, an average of 1 year
  Quantitative Indicators，the maximum area bounded by the luminal border on OCT
Percent area stenosis | through study completion, an average of 1 year
  Quantitative Indicators，the (reference lumen area minus the minimum lumen area) divided by the reference lumen area, multiplied by 100. The reference segment used should be specified (proximal, distal, largest or average) on OCT
Mean stent area | through study completion, an average of 1 year
  Quantitative Indicators，the mean area bounded by the stent border on OCT
Minimum stent area | through study completion, an average of 1 year
  Quantitative Indicators，the Minimum area bounded by the stent border on OCT
Maximum stent area | through study completion, an average of 1 year
  Quantitative Indicators，the Maximum area bounded by the stent border on OCT
lipid-laden intima | through study completion, an average of 1 year
  Qualitative indicators,a diffusely bordered, signal-poor region with overlying signal-rich bands in the intima on OCT.the investigators measured its incidence on OCT.
Calcification | through study completion, an average of 1 year
  Qualitative indicators,shows a well-delineated, signal-poor region with sharp borders.the investigators measured its incidence on OCT.
Thrombi | through study completion, an average of 1 year
  Qualitative indicators,masses protruding into the lumen and discontinuous from the surface of the vessel wall.the investigators measured its incidence on OCT.
Intimal rupture | through study completion, an average of 1 year
  Qualitative indicators,discontinuity of the fibrous cap connecting the lumen.the investigators measured its incidence on OCT.
Neovascularization | through study completion, an average of 1 year
  Qualitative indicators,the presence of signal-poor holes or tubular structures with a diameter of 50 to 300 μm that are not connected to the vessel lumen.the investigators measured its incidence on OCT.
Thin-cap fibroatheroma (TCFA) | through study completion, an average of 1 year
  containing intima was defined as fibrous cap thickness ≤65 μm at the thinnest segment and an angle of lipid tissue ≥180°.the investigators measured its incidence on OCT.
Macrophage infiltration | through study completion, an average of 1 year
  Qualitative indicators,a bright spot with a high signal variance from the surrounding tissue.the investigators measured its incidence on OCT.
Stent underexpansion | through study completion, an average of 1 year
  Qualitative indicators,Stent expansion describes the minimum stent cross-sectional area either as an absolute measure (absolute expansion), or compared with the predefined reference area, which can be the proximal, distal, largest, or average reference area (relative expansion).the investigators measured its incidence on OCT.
stent fracture | through study completion, an average of 1 year
  Qualitative indicators,the interruption of stent continuity.the investigators measured its incidence on OCT.
Uncovered struts | through study completion, an average of 1 year
  the ratio of uncovered-to-total stent struts per section was calculated and expressed as percent on OCT.
neoatherosclerosis | through study completion, an average of 1 year
  neoatherosclerosis were defined by the presence of one or more of the following: lipid laden tissue ，thin-cap fibroatheroma (TCFA)，neointimal calcification，Macrophage infiltration.the investigators measured its incidence .

CONTACTS AND LOCATIONS:
Overall Officials: geng wang, M.D., Study Chair — The General Hospital of Northern Theater Command
Locations (1):
- ShenyangNH, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided
The provision of individual patient data requires the informed consent of the patient. In addition, basic information about the patient and coronary angiography results may be provided in the form of pictures or videos. OCT results need to be analyzed in specialized offline software, and the investigators provide the most intuitive OCT results possible.